CLINICAL TRIAL: NCT01203436
Title: Supplemental Therapeutic Oxygen for Prethreshold Retinopathy of Prematurity
Acronym: STOP-ROP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Eye Institute (NEI) (NIH); National Institute of Nursing Research (NINR) (NIH); Delta Gamma Sorority (Unknown); Rhea and Raymond White (Unknown); Research to Prevent Blindness (Other)
Responsible Party: Dale L. Phelps/ Lead Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0010; U10HD027904 (NIH); U10HD027851 (NIH); U10HD027856 (NIH); U10HD027880 (NIH); U10HD027853 (NIH); U10HD021415 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); M01RR000054 (NIH); M01RR000070 (NIH); NCT00000141 (obsolete NCT alias)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Retinopathy of Prematurity; Blindness
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity; Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental Oxygen (Experimental): Supplemental oxygen to achieve a pulse oximetry target range of 96% to 99%.
  Interventions: Procedure: Supplemental Oxygen Management
- Conventional Oxygen (Active Comparator): Conventional oxygenation at a pulse oximetry target of 89% to 94%.
  Interventions: Procedure: Conventional Oxygen Management

INTERVENTIONS:
Procedure: Supplemental Oxygen Management — Supplemental arm with pulse oximetry targeted at 96% to 99% saturation, for at least 2 weeks, and until both eyes were at study endpoints.
  Arms: Supplemental Oxygen
Procedure: Conventional Oxygen Management — Conventional oxygen arm with pulse oximetry targeted at 89% to 94% saturation.
  Arms: Conventional Oxygen

SUMMARY:
The purpose of this trial was to determine the efficacy and safety of supplemental therapeutic oxygen for infants with prethreshold retinopathy of prematurity (ROP) to reduce the probability of progression to threshold ROP and the need for peripheral retinal ablation.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is an abnormal growth of the blood vessels in the eye that occurs primarily in very premature infants. Eye development occurs normally in the womb; in infants born prematurely, however, the blood vessels must finish developing outside the protective environment of the uterus. Retinopathy of prematurity (also known as retrolental fibroplasia) is a leading cause of blindness and other vision impairments (myopia, strabismus, and amblyopia) in children, both in developed and developing countries.

This study was a randomized trial comparing the effects of 2 oxygenation strategies on the progression of ROP. Infants with prethreshold ROP in at least one eye were eligible for the study. Enrolled infants were randomized to receive either conventional oxygenation at a pulse oximetry target of 89% to 94%, or supplemental oxygen to achieve a pulse oximetry target range of 96% to 99%. Infant were placed on continuous pulse oximetry monitoring and to maintain oxygen saturation, as much as possible, in the assigned target range.

ELIGIBILITY:
Inclusion Criteria:

* Infants with prethreshold retinopathy of prematurity, confirmed by 2 certified ophthalmologic exams
* Median pulse oxygen saturation <94% in room air
* Median pulse oxygen saturation can be kept safely >96% on oxygen/ventilator

Exclusion Criteria:

* No fatal congenital anomaly or congenital eye anomaly

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 649 (Actual)
Dates: Start 1994-02; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Progression from moderate to severe ROP (prethreshold) to threshold ROP requiring peripheral ablative surgery | 3 months of age
  Progressing from moderate ROP (prethreshold) to threshold ROP requiring peripheral ablative surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dale L. Phelps, MD, Study Director — University of Rochester; Neal L. Oden, PhD, Principal Investigator — The Emmes Company, LLC; Cynthia Cole, MD, Principal Investigator — Tufts Medical Center; Richard E. McClead, MD, Principal Investigator — Ohio State University; Alan R. Spitzer, MD, Study Director — Thomas Jefferson University; J. David Bradford, MD, Principal Investigator — Arkansas Childrens Hospital; Charles C. Barr, MD, Principal Investigator — University of Louisville; William Oh, MD, Principal Investigator — Brown University, Womens and Infants Hospital; Barbara J. Stoll, MD, Principal Investigator — Emory University; James A. Lemons, MD, Principal Investigator — Indiana University; David K. Stevenson, MD, Principal Investigator — Stanford University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee at Memphis; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; David Easa, MD, Principal Investigator — Kapiolani Medical Center; Beverly S. Brozanski, MD, Principal Investigator — Magee-Womena Hospital; Robert Gordon, MD, Principal Investigator — Tulane University; Pamela A. Weber, MD, Principal Investigator — SUNY Stonybrook; Frank W. Kokomoor, MD, Principal Investigator — Akron Childrens Hospital; Michael J. Shapiro, MD, Principal Investigator — University of Illinois at Chicago; Raul C. Banagale, MD, Principal Investigator — Legacy Emanual Childrens Hospital; Mitchell E. Stern, MD, Principal Investigator — Sheridan Childrens Healthcare Services; Mark W. Preslan, MD, Principal Investigator — University of Maryland; Shephen S. Feman, MD, Principal Investigator — Vanderbilt University; James Kirk, DO, Principal Investigator — University of Florida; Terri L. Young, MD, Principal Investigator — Fairview University Medical Center; Mary Anne McCaffree, MD, Principal Investigator — Childrens Hospital of Oklahoma; Malini Satish, MD, Principal Investigator — Childrens Medical Center of Northwest Ohio; Patrick J. Droste, MD, Principal Investigator — Cook Institute for Research and Education
Locations (9):
- United States (9):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Supplemental Therapeutic Oxygen for Prethreshold Retinopathy Of Prematurity (STOP-ROP), a randomized, controlled trial. I: primary outcomes. Pediatrics. 2000 Feb;105(2):295-310. doi: 10.1542/peds.105.2.295. PMID 10654946
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/